CLINICAL TRIAL: NCT04703231
Title: Comparison of Ocular Findings in Patients Between Surgical and Natural Menopause
Status: Completed | Type: Observational
Sponsor: Batman Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erhan Okuyan,M.D, Principle investigator, Batman Training and Research Hospital
Other Study IDs: 20201987
Record Dates: First submitted 2021-01-01; First posted 2021-01-11 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Menopause Surgical; Macula Edema; Visual Acuity Reduced Transiently
Keywords: menopause; Eye disease; Macular changes
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Natural menopause(Control group): Female patients between 45-60 years of age diagnosed with menopause without any intervention
  Interventions: Diagnostic Test: measurement of macular thickness, corneal thickness and lens opacities
- Surgical Menopause (Case group): Female patients aged 45-60 years included in the study 3 months after bilateral oophorectomy and hysterectomy
  Interventions: Diagnostic Test: measurement of macular thickness, corneal thickness and lens opacities

INTERVENTIONS:
Diagnostic Test: measurement of macular thickness, corneal thickness and lens opacities — The incidence of macular thickness, Corneal thickness, intraocular pressure and lens opacities will be investigated by an ophthalmologist.

SUMMARY:
It is aimed to compare the ocular findings in patients with natural and surgical menopause.

DETAILED DESCRIPTION:
To compare the parameters such as fundus examination, macular thickness, visual acuity and lens opacities among female patients diagnosed with menopause between the ages of 40-65.The criteria for exclusion from the study are the presence of a history of illness, drug use, smoking and alcohol use.Inclusion criteria were female patients who were in menopause and who did not use any medications. For surgical menopause, the uterus and ovaries were surgically removed at least 3 months ago.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed menopause (Natural or Surgical Menopause( At least 3 months after surgery),
* No history of illness(Diabetes,Heart disease,Kidney disease etc.)
* Not Smoking
* Did not use alcohol
* Have not use any medication
* Age between 45-65 years
* BMI between 20-25 kg/m

Exclusion Criteria:

* Smoking or Alchohol consumption
* Age before 45 and after 65 years
* Have chronic disease
* Using any medication
* Have not diagnosed Menopause
* BMI greater than 30 kg/m

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Will be studied in a patient population with low sociocultural level.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Macular thickness measurement | 3 months after menopause
  Macular thickness(micron) in both eyes will be measured by optical coherence tomography,
Detecting lens opacities | 3 months after menopause
  Lens opacities (Grade 1,2,3,4) will be measured by indirect biomicroscopy,
Intraocular pressure measurement | 3 months after menopause
  Intraocular pressures( mm Hg) will be measured and recorded with the applanation tonometry device.
Comparison of all detected data | 3 months after menopause
  All numerical data will be analyzed and compared with relevant statistical tests and the p value will be accepted as less than 0.05 to be considered a statistically significant difference.

CONTACTS AND LOCATIONS:
Locations (1):
- Batman Maternity and Child Health Hospital, Batman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No